CLINICAL TRIAL: NCT04445389
Title: A Phase 1/2a, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Immunogenicity of GX-19, a COVID-19 Preventive DNA Vaccine in Healthy Subjects
Brief Title: Safety and Immunogenicity Study of GX-19, a COVID-19 Preventive DNA Vaccine in Healthy Adults
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to change the investigational product for a strategic reason.
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: GX-19-HV-001
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase 1: Open-label, Dose escalation (3-arms) Phase 2a: Randomized, Double-blinded, Placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GX-19: Dose A (Experimental): Dose A of GX-19 will be intramusculary administered via EP on day 1 and day 29.
  Interventions: Drug: GX-19
- GX-19: Dose B (Experimental): Dose B of GX-19 will be intramusculary administered via EP on day 1 and day 29.
  Interventions: Drug: GX-19
- GX-19: Dose C (Placebo Comparator): Dose C of GX-19 will be intramusculary administered via PharmaJet® Needle Free Delivery on day 1 and day 29.
  Interventions: Drug: GX-19
- Placebo: Dose A, B, or C (Placebo Comparator): Placebo will be intramusculary administered on day 1 and day 29 via EP or PharmaJet® Needle Free Delivery
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: GX-19 — DNA vaccine expressing SARS-CoV-2 S-protein antigen
  Other Names: DNA vaccine expressing SARS-CoV-2 S-protein antigen
  Arms: GX-19: Dose A; GX-19: Dose B; GX-19: Dose C
Drug: Saline — Saline
  Arms: Placebo: Dose A, B, or C

SUMMARY:
The objective of our study is to evaluate safety, tolerability, and immunogenicity of COVID-19 preventive DNA vaccine in healthy volunteers.

DETAILED DESCRIPTION:
This clinical study is phase 1/2a clinical trial to evaluate safety, tolerability, and immunogenicity of COVID-19 preventive vaccine by intramuscularly administration in healthy volunteers.

Phase 1 of this study is designed as dose escaltion, single arm, open-labeled and a total of 60 subjects will be enrolled. Phase 2a of study is designed as randomized, double-blind, placebo controlled and a total of 150 subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following criteria during the screening period:

1. Able and willing to comply with all study procedures and voluntarily signs informed consent form
2. Healthy adult male or female aged 19-50 years
3. Those who weigh 50 kg to 90kg and have a body mass index (BMI) of 18.0 kg/m2 to 28.0 kg/m2 at screening visit.
4. Willing to provide specimens such as blood and urine during the study, including end of study visit.

Exclusion Criteria:

Participants meeting any of the following criteria at the Screening Visit:

1. Immunosuppresion including immunodeficiency disease or family history
2. Any history of malignant disease within the past 5 years
3. Scheduled to undergo any surgery or dental treatment during the study
4. Having received immunoglobulin or blood-derived drugs or being expected to be administered within 3 months prior to administration.
5. Having relied on antipsychotic drugs and narcotic analgesics within 6 months before administration
6. Positive of serum test at screening
7. Suspected of drug abuse or a history within 12 months prior to administration
8. Active alcohol use or history of alcohol abuse
9. Serious adverse reaction to a drug containing GX-19 or other ingredients of the same categories or to a vaccine or antibiotic, nonsteroidal anti-inflammatory disease control, etc. or an allergic history
10. History of hypersensitivity to vaccination such as Guillain-Barre syndrome
11. Those who have or with a history of disease corresponding to other hepatobiliary, kidneys, nervous systems (middle or peripheral), respiratory machines (e.g. asthma, pneumonia, etc., endocrine systems (uncontrolled diabetes, hyperlipidemia, etc.) and cardiovascular (congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension), blood tumors, urinary machines, mental, musculoskeletal systems, immune system (rheumatoid arthritis, systemic arthritis, mumps, immunodeficiency disease)
12. Having hemophilia at risk of causing serious bleeding when injected intramuscularly or receiving anticoagulants
13. Subjects who have been contact with COVID-19 infections in the past prior to administration, have been classified as COVID-19 confirmed patients, medical patients or patients with symptoms or have been identified with SARS and MERS infection history in the past
14. Acute fever, cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to administration
15. Other vaccination history within 28 days prior to the administration or being scheduled to be inoculated during the study
16. History of having taken immunosuppressant or Immune modifying drug within 3 months prior to administration
17. Having participated and had clinical trial drug administration in another clinical trial or biological equivalence study within 6 months prior to the administration
18. Pregnant or breastfeeding female, however, those are allowed to participate in the study only if they stop breastfeeding before participation (fertile female† must be negative in serum pregnancy test at screening
19. Fertile female who do not agree to use effective contraception methods (condoms, contraceptive diaphragm, intrauterine contraceptive devices) during the study
20. Any other clinically significant medical or psychiatric finding which is considered inappropriate by investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events | Through 1 year post vaccination
  solicited local and systemic AEs after vaccination
Incidence of unsolicited adverse events | Through 1 year post vaccination
  unsolicited AEs after vaccination
Incidence of serious adverse events | Through 1 year post vaccination
  percentage of subjects with SAEs

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of antigen-specific binding antibody titers | Through 1 year post vaccination
  Change from baseline in antigen-specific binding antibody titers
Percentage of subjects who seroconverted after vaccination | Through 1 year post vaccination
  Seroconversion rate can be calculated based on test results reaching the quantifiable antibody level after vaccination
Geometric mean titer (GMT) of neutralizing antibody level | Through 1 year post vaccination
  NAb is regarded as produced when FRNT50 is detected more than four times the baseline after vaccination
Geometric mean fold rise (GMFR) of antigen-specific binding antibody titers | Through 1 year post vaccination
  Change from baseline in antigen-specific binding antibody titers

OTHER OUTCOMES:
Change from baseline in antigen-specific IFN-g cellular immune response | Through 1 year post vaccination
  Antigen-specific IFN-γ T cell immune response assessed before/after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: JungWon Woo, Ph.D., Study Director — Genexine, Inc.
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No